CLINICAL TRIAL: NCT00274287
Title: A Phase II Pilot Study Investigating the Efficacy and Activity of Single Agent GM-CSF (Leukine) Maintenance Approach in Androgen-independent Prostate Cancer (AIPC) Patients Responding to Taxotere Chemotherapy
Brief Title: GM-CSF for Maintenance of Prostate Cancer for Patients Responding to Taxotere
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oncology Specialists, S.C. (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, Dr. Sigrun Hallmeyer, Principal Investigator, Oncology Specialists, S.C.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0412; NCT00336037 (obsolete NCT alias)
Record Dates: First submitted 2006-01-06; First posted 2006-01-10 (Estimated); Results first posted 2012-05-09 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Colony-Stimulating Factors; sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GM-CSF (Experimental): Once patients have finished receiving the chemotherapy and no signs of disease progression they may receive GM-CSF as outlined in the protocol
  Interventions: Drug: GM CSF

INTERVENTIONS:
Drug: GM CSF — 250 ug/m2 daily for 2 weeks followed by 2 weeks of rest
  Other Names: Leukine

SUMMARY:
This trial is designed to investigate the efficacy and safety of GM-CSF used as a maintenance program in patients with androgen-independent prostate cancer (AIPC) who have achieved a maximal response on a taxotere or other chemotherapy schedule.

DETAILED DESCRIPTION:
Patients will be treated on this single arm, open label trial until primary end point is met, patient's withdrawal, or investigator's discretion. After achieving a maximal response on taxotere or other chemo schedule they were eligible to enroll in this trial and begin treatment with maintenance GMCSF for 2 weeks followed by 2 weeks of rest. Once progression was documented the patients were taken off study.

ELIGIBILITY:
Inclusion Criteria:

1. Men >18 years of age. No upper age limit
2. Written informed consent approved by institutional review board should be explained to and signed by patient
3. Documentation of histologically confirmed adenocarcinoma of the prostate. Gleason score of any sum is allowed on this study.
4. Metastatic disease as evidenced by visceral involvement, bone disease, or PSA elevation.
5. Patients should meet the criteria of androgen independent prostate cancer (AIPC). Patients would fulfill these criteria if they continue to progress despite complete androgen blockade (surgical or medical castration with anti-androgen) and despite an anti-androgen withdrawal trial. Failing anti-androgen withdrawal is defined as no decline by 25% or more 3-weeks after stopping anti-androgens.

   Progression on hormonal therapy is defined as ANY of the following:
   * PSA: 2 consecutive rising PSA values, at least 14-days apart, each being > 5 ng/ml
   * For patients with visceral measurable disease, progression is defined as an increase by 50% or more in the size of measurable areas, or any development of new lesions.
   * For patients with bone-only disease, progression is defined as the appearance of 2 or more new areas of abnormal uptake on a bone scan, when compared to prior imaging studies. Changes in the uptake of already existing lesions will NOT be used to define progressive disease.
   * For patients with bone AND visceral disease, fulfilling any of the criteria in 5.2 or 5.3 is sufficient to define progression.
6. Castration levels of testosterone (< 50 ng/dl) achieved via medical or surgical castration. Patients should continue on LHRH agonists throughout if this is the method used to achieve castration.
7. Life expectancy of at least 6 months
8. Adequate hematologic, renal, and liver function as evidenced by the following:

   * WBC > 2000,
   * ANC > 1000,
   * Platelet count > 100,000,
   * HgB > 9.0 g/dl, Creatinine < 2,
   * Total bilirubin < 2x upper limit of normal,
   * AST and ALT < 3 x upper limit of normal
9. ECOG performance status of 0 or 1.
10. The use of intravenous polyphosphates for bone metastases is allowed.
11. upon completion of the taxotere portion of study, patient can be enrolled & receive GM-CSF if ANY of the following criteria is met:

    * Patients received total of 8 cycles of taxotere & have no signs of disease progression
    * Patients achieved their maximal response despite receiving < than 8 cycles of taxotere. Maximum response is defined as a drop in measures of PSA by 10% or less on 2 consecutive measurements.
    * Patients who have completed their chemotherapy < than 12 weeks prior to opening this trial & still have stable disease without progression (by PSA and radiographically) will be eligible to receive maintenance GM-CSF

Exclusion Criteria:

1. presence of brain metastases
2. Known HIV+ status
3. ECOG performance status of 2 or higher
4. Use of investigational agents within 4 weeks of starting
5. Patients with prior exposure to more than one chemotherapy program Patients who have received one chemotherapy schedule can be enrolled on study and receive GM-CSF (the maintenance arm) if their last chemotherapy was taxotere, given within the past 12 weeks, and they have demonstrated NO evidence of progression radiographically and biochemically. Prior exposure to steroids is NOT an exclusion criteria.
6. Patients with other active malignancies (excluding non-melanoma skin cancers)are excluded. Prior malignancies are not exclusion criteria as long as last treatment for such malignancies was over 5 years prior to enrollment.
7. Treatment with investigational products are NOT an exclusion criteria, if therapy was last received over 4 weeks prior to enrollment.
8. Any medical intervention or other condition which, in the opinion of the principle investigator, could compromise adherence with study requirements.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chadi Nabhan, MD, Principal Investigator — Oncology Specialists, SC
Locations (1):
- Oncology Specialists, SC, Park Ridge, Illinois, United States

REFERENCES:
- [Result] Nabhan C, Meyer A, Tolzien K, Bitran JD, Lestingi TM. A phase II pilot trial investigating the efficacy and activity of single agent granulocyte macrophage colony-stimulating factor as maintenance approach in castration - resistant prostate cancer patients responding to chemotherapy. Avicenna J Med. 2011 Jul;1(1):12-7. doi: 10.4103/2231-0770.83718. PMID 23210004

RESULTS

PARTICIPANT FLOW:
Groups:
- GM-CSF (Leukine): Once patients have finished receiving the chemotherapy and no signs of disease progression they may receive GMCSF (Leukine) as outlined in the protocol. 250 micro grams/m2 daily for two weeks followed by two weeks of rest.
Period: Overall Study
Arm/Group | GM-CSF (Leukine)
Started | 15
Completed | 13
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — subject non-compliance | 1

BASELINE CHARACTERISTICS:
Arm/Group | GM-CSF (Leukine)
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] — Age at protocol entry
  years | 78 [66 to 96]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15
Gleason Score >=7 [Count of Participants; unit: Participants] — the Gleason score is used to help evaluate the prognosis of men with prostate cancer. A Gleason score is given to prostate cancer based upon its microscopic appearance. Cancers with a higher Gleason are more aggressive and have a worse prognosis. Scores range from 2-10.
  Participants | 14
Median time from diagnosis to GM-CSF [Median (Full Range); unit: months] — granulocyte macrophage colony-stimulating factor
  months | 71 [19 to 145]
Median number of prior therapies [Median (Full Range); unit: therapies] | 2 [1 to 3]
median PSA [Median (Full Range); unit: ng/dl] | 51.7 [0.1 to 566]
Median alkphos [Median (Full Range); unit: U/L] | 97 [31 to 245]
Prior initial therapy [Count of Participants; unit: Participants]
  RT (radiation therapy) | 5
  ADT (androgen deprivation therapy) | 7
  RP (radical prostatectomy) | 3
Site of Metastases [Count of Participants; unit: Participants]
  bone | 7
  visceral disease | 1
  viseral and bone | 7

OUTCOME MEASURES:

1. Primary Outcome: Time to Disease Progression (TTP)
Description: The primary end point of this study is to evaluate time to disease progression (TTP). TTP is defined as the time from starting taxotere until there is evidence of progressive disease (PD) as defined below (radiographically and/or biochemically). PD was defined as more than 20% in the sum of longest diameter of measurable lesions compared to baseline, and/or evidence of new lesions on imaging studies. Median TTP from GM-CSF administration and Median TTP from start of chemotherapy is being reported
Time Frame: up to 21 months
Population: all evaluable participants
Measure: Median (Full Range); unit: months
Groups:
- GM-CSF (Leukine): Taxotere is given at 75 mg/m2 on day 1 intravenously over 60 minutes with appropriate and standard pre-medications. Patients are eligible to receive growth factor support with G-CSF or Neulasta on day 2 at the investigator's discretion.
Arm/Group | GM-CSF (Leukine)
Number analyzed (Participants) | 13
months
  TTP from GM-CSF | 6 [2 to 12]
  TTP from chemotherapy | 11 [9 to 21]

2. Secondary Outcome: Response Rate (PSA)
Description: Biochemical PR (Partial Response) was defined as a PSA that decreases by 50% and maintains by at least 3 weeks by confirmatory measurement. Biochemical SD (stable disease) was defined as a PSA that was increased by less than 25% or decreased by less than 50% Biochemical PD (progressive disease) was defined as an increase of at least 25% confirmed 3 weeks after.
Time Frame: up to 21 months
Population: all evaluable participants
Measure: Count of Participants; unit: Participants
Arm/Group | GM-CSF (Leukine)
Number analyzed (Participants) | 13
Participants
  PSA PD | 7
  PSA PR | 2
  PSA SD | 4

3. Secondary Outcome: Response Rate (Radiographic)
Description: PR was defined as more than 30% decrease in the sum of the longest diameter of measurable lesions compared to baseline. SD was defined when lesions did not meet criteria for PR or PD. PD was defined as more than 20% increase in the sum of the longest diameter of measurable lesions compared to baseline, and/or evidence of new lesions at imaging studies. The appearance of 2 or more new boney lesions on bone scan development of cord compression, and pathologic fractures constituted PD.
Time Frame: up to 21 months
Population: all evaluable participants
Measure: Count of Participants; unit: Participants
Arm/Group | GM-CSF (Leukine)
Number analyzed (Participants) | 13
Participants
  Radiographic PD | 4
  Radiographic SD | 9

4. Secondary Outcome: Median Overall Survival (OS)
Time Frame: up to 44 months
Population: all evaluable participants
Measure: Median (Full Range); unit: months
Arm/Group | GM-CSF (Leukine)
Number analyzed (Participants) | 13
months
  OS from GM-CSF | 12 [2 to 38]
  OS from chemotherapy | 21 [10 to 44]

5. Secondary Outcome: Median Number of GM-CSF Cycles
Time Frame: up to 12 months
Population: all evaluable participants
Measure: Median (Full Range); unit: months
Arm/Group | GM-CSF (Leukine)
Number analyzed (Participants) | 13
months | 6 [2 to 12]

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | GM-CSF (Leukine)
Serious Adverse Events (participants affected / at risk) | 7/15
Other Adverse Events (participants affected / at risk) | 7/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GM-CSF (Leukine) (N=15)
Angina (Cardiac disorders) | 1 (2)
edema (Vascular disorders) | 1 (1)
dehydration (General disorders) | 1 (2)
pnuemonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
weakness (General disorders) | 2 (2)
meningioma (General disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 1 (1)
dizziness (General disorders) | 1 (1)
bowel obstruction (Gastrointestinal disorders) | 1 (3)
Anemia (Blood and lymphatic system disorders) | 1 (1)
A Fib (Cardiac disorders) | 1 (1)
Port infection (General disorders) | 2 (2)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
syncope (General disorders) | 2 (2)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Thrush (Infections and infestations) | 1 (1)
DVT (Vascular disorders) | 1 (1)
fatigue (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GM-CSF (Leukine) (N=15)
albumin low (Blood and lymphatic system disorders) | 6 (6)
alk phos (Blood and lymphatic system disorders) | 4 (4)
alopecia (General disorders) | 3 (3)
anorexia (Metabolism and nutrition disorders) | 4 (4)
arthralgia (Surgical and medical procedures) | 1 (1)
AST high (Hepatobiliary disorders) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
balance difficulty (Nervous system disorders) | 1 (1)
bleeding (Blood and lymphatic system disorders) | 2 (2)
breathing difficult (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bruising (Blood and lymphatic system disorders) | 2 (2)
BUN (Hepatobiliary disorders) | 3 (3)
Calcium low (Blood and lymphatic system disorders) | 6 (6)
Carbon Dioxide (Respiratory, thoracic and mediastinal disorders) | 2 (2)
cellulitis (Musculoskeletal and connective tissue disorders) | 1 (1)
chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
chills (General disorders) | 3 (3)
chloride low (Blood and lymphatic system disorders) | 2 (2)
chloride high (Blood and lymphatic system disorders) | 1 (1)
concentration difficulty (Nervous system disorders) | 1 (1)
confusion (Nervous system disorders) | 1 (1)
conjunctiva abnormal (Eye disorders) | 1 (1)
constipation (Gastrointestinal disorders) | 5 (5)
cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
creatinine low (Blood and lymphatic system disorders) | 1 (1)
depression (Psychiatric disorders) | 2 (2)
disoriented (Nervous system disorders) | 1 (1)
DOE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
dysphasia (Nervous system disorders) | 1 (1)
E coli (Infections and infestations) | 1 (1)
ear pain (Ear and labyrinth disorders) | 2 (2)
eyes dry (Eye disorders) | 1 (1)
eyes watery (Eye disorders) | 1 (1)
fall (Nervous system disorders) | 2 (2)
fever (Infections and infestations) | 3 (3)
headache (Nervous system disorders) | 1 (1)
heart beat rapid (Cardiac disorders) | 3 (3)
hives (General disorders) | 1 (1)
HOH (Ear and labyrinth disorders) | 1 (1)
hot flashes (Endocrine disorders) | 2 (2)
hyperglycemia (Endocrine disorders) | 3 (3)
hyperlipedmia (Blood and lymphatic system disorders) | 1 (1)
hypertension (Cardiac disorders) | 1 (1)
hyponatremia (Blood and lymphatic system disorders) | 6 (6)
incontinence (Renal and urinary disorders) | 1 (1)
insomnia (General disorders) | 2 (2)
itching (Skin and subcutaneous tissue disorders) | 2 (2)
leg ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
libido decreased (General disorders) | 1 (1)
lightheadedness (Nervous system disorders) | 1 (1)
lymphopenia (Blood and lymphatic system disorders) | 1 (1)
memory loss (Nervous system disorders) | 2 (2)
mouth dryness (General disorders) | 2 (2)
mouth sores (Skin and subcutaneous tissue disorders) | 1 (1)
nail changes (Skin and subcutaneous tissue disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 7 (7)
neuralgia (Nervous system disorders) | 2 (2)
nocturia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pain (General disorders) | 5 (5)
phosporus low (Blood and lymphatic system disorders) | 1 (1)
potassium low (Blood and lymphatic system disorders) | 1 (1)
protein low (Gastrointestinal disorders) | 5 (5)
rash (Skin and subcutaneous tissue disorders) | 5 (5)
redness (Skin and subcutaneous tissue disorders) | 1 (1)
seeing difficulties (Eye disorders) | 6 (6)
seizure (Nervous system disorders) | 1 (1)
sinus problems (Respiratory, thoracic and mediastinal disorders) | 1 (1)
skin dry (Skin and subcutaneous tissue disorders) | 2 (2)
sore throat (Infections and infestations) | 3 (3)
swallowing difficulty (Gastrointestinal disorders) | 1 (1)
swelling (Blood and lymphatic system disorders) | 2 (2)
sweats (General disorders) | 3 (3)
thrombocytopenia (Blood and lymphatic system disorders) | 3 (3)
urination problems (Renal and urinary disorders) | 2 (2)
urinary retention (Renal and urinary disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 4 (4)
weight loss (Gastrointestinal disorders) | 6 (6)
welts (Skin and subcutaneous tissue disorders) | 1 (1)
wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
CAD (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less